CLINICAL TRIAL: NCT05928676
Title: Effects of S-allylcysteine-rich Garlic Extract and Dietary Inorganic Nitrate Formula (Vascanox® HP) on Blood Pressure and Nitric Oxide Levels: an Open-label Clinical Trial Among Hypertensive Adults
Brief Title: Open Label Clinical Trial of Vascanox® HP on Nitric Oxide and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calroy Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 022-CalroyHS
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-06

CONDITIONS: Hypertension; Elevated Blood Pressure
Keywords: hypertension; elevated blood pressure; nitric oxide; S-allylcysteine; dietary nitrate; Vascanox HP
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vascanox® HP (Experimental)
  Interventions: Dietary Supplement: Vascanox® HP

INTERVENTIONS:
Dietary Supplement: Vascanox® HP — Vascanox® HP is a proprietary formulation that combines dietary sources of nitric oxide and hydrogen sulfide aimed at increasing the levels and duration of nitric oxide biosynthesis. Vascanox® HP contains an advanced blend of berry extracts in addition to beet root powder, black garlic, vitamin C, and minerals known to influence nitric oxide biosynthesis and metabolism. Because of the particular combination of ingredients, Vascanox® HP is expected to affect both canonical and non-canonical pathways of nitric oxide production and to augment nitric oxide reservoir in the body leading to an increased and prolonged nitric oxide bioavailability.

SUMMARY:
Conversion of dietary nitrates to nitric oxide (NO) is a non-canonical pathway that plays an important role in NO biology, particulalry under pathological conditions. Nitrate supplementation has been shown to help control mild hypertension. Recent studies have suggested that another gaseous transmitter, hydrogen sulfide, also influences NO biosynthesis and metabolism. This open-label clinical trial will evalute the effect of Vascanox® HP, a proprietary formulation that combines dietary sources of nitric oxide and hydrogen sulfide, on nitric oxide bioavailability and on blood pressure in subjects experiencing elevated blood pressure. Participants will supplement with Vascanox® HP for four weeks. Blood pressure will be measured at baseline, two weeks, and fours weeks. Salivary nitric oxide will be assessed prior to and two, six, and 24 hours after dosing on the first day of the study and prior to and two hours after dosing at subsequent study visits. Participants will also self-monitor their saliva nitric oxide levels and blood pressure daily for 4 weeks. Changes in study outcomes over time will be evaluated via analysis of variance (ANOVA) and paired t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Mild hypertension defined as brachial artery blood pressure greater than or equal to 130 mm Hg systolic and less than or equal to 140 mm Hg systolic or greater than or equal to 85 mm Hg diastolic or less than 90 mm Hg diastolic while taking or not taking antihypertensive drugs.
* Not currently taking nitric oxide supplements, and not consuming nitric oxide supplements for 14 days prior to screening.
* Ability to give written informed consent.
* Ability to adhere to study protocol directives and procedures.

Exclusion Criteria:

* Initiated or had a dose change of an antihypertensive agent less than 6 months prior to the enrollment date.
* A positive nitric oxide saliva test strip (result >2) on the day of Screening.
* A positive nitric oxide saliva test strip (result >2) on the day of Baseline/Visit 1.
* A high saliva NO3 test strip result (result >2) but a low NO test strip result.
* Current use of antibiotics.
* Chronic steroid use >15 mg daily.
* Previous myocardial infarction less than 2 years of enrollment date.
* Unstable angina.
* Previous stroke or transient ischemic attack (TIA) less than 2 years of enrollment date.
* Uncompensated congestive heart failure (CHF).
* Previous percutaneous transluminal coronary angioplasty (PTCA) or stent less than 2 years of enrollment date.
* Previous coronary arterial bypass graft (CABG) less than 2 years of enrollment date.
* Known or previous cancer less than 5 years of enrollment date.
* Type 1 diabetes mellitus.
* Prescribed dosing with insulin, injectable or inhaled.
* Pregnant females.
* Females of child bearing age not on an accepted contraception control method.
* Allergy/sensitivity to study products or their ingredients.
* Current drug or alcohol use or dependence that, in the opinion of the principal investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual to give written informed consent.
* Current or past participation within 30 calendar days in another clinical trial, as warranted by the administration of this intervention.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-24 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Assessed at baseline, at 2 weeks, and at the 4 week conclusion of study
  Change in blood pressure in millimeters of mercury (mmHg) assessed in the branchial artery

SECONDARY OUTCOMES:
Salivary nitric oxide | Salivary nitric oxide assessed prior to and two hours after dosing at baseline, 2 weeks, and at the 4 week conclusion of the study. Salivary nitric oxide will be additionally assessed at 6 and 24 hours after dosing on the first day of the study only.
  Salivary levels of nitric oxide assessed using commercially available FDA registered strips. Nitric oxide test strips measure nitrite, which is used as an established surrogate marker for nitric oxide.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Houston, M.D., Principal Investigator — The Hypertension Institute
Locations (1):
- The Hypertension Institute, Nashville, Tennessee, United States